CLINICAL TRIAL: NCT04019782
Title: Efficacy Evaluation of Intraarticular Collagen-polyvinyl Pyrrolidone (Fibroquel®) vs Hylan G-F 20 (Synvisc®) in the Treatment of Knee Osteoarthritis. A Double-blind, Controlled, Randomised, Parallel-group Non-inferiority Study
Brief Title: Collagen-PVP vs Hylan G-F 20 in the Treatment of Knee Osteoarthritis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R-2018-785-041
Record Dates: First submitted 2019-07-11; First posted 2019-07-15 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Knee Osteoarthritis; Gonarthrosis
Keywords: Osteoarthritis; Intraarticular Injections; Viscosupplementations; Type I Collagen; Patient Outcome Assessment; Patient Reported Outcome Measures
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Osteogenesis Imperfecta, Type IV | interventions — collagen-PVP

STUDY DESIGN:
Intervention Model Description: Participants in one group receive drug A (Hylan G-F20) "in parallel" to participants in the other group, who receive drug B (Collagen-PVP).
Who Masked: Participant, Outcomes Assessor
Masking Description: Double-blind masking.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Collagen-PVP (Experimental): Collagen-polyvinyl pyrrolidone (collagen-PVP).
  Interventions: Drug: Collagen-PVP
- Hylan G-F 20 (Active Comparator): Hylan G-F 20.
  Interventions: Device: Hylan G-F 20

INTERVENTIONS:
Drug: Collagen-PVP — Infiltrations of 1.5 ml collagen-polyvinyl pyrrolidone (collagen-PVP) plus 1 mL of 2% xylocaine without epinephrine, administered by intraarticular injections (three doses, one each 7 days)
  Other Names: Fibroquel
  Arms: Collagen-PVP
Device: Hylan G-F 20 — Infiltrations of 2 mL 0.8% Hylan G-F 20 (16 mg) solution, administered by intraarticular injections (three doses, one each 7 days)
  Other Names: Synvisc
  Arms: Hylan G-F 20

SUMMARY:
Articular cartilage degradation is the main characteristic of osteoarthritis (OA), involving enzymatic and inflammatory mechanisms that change it into a chronic disease. Since articular cartilage shows limited regenerative ability, several intra-articular drugs have been developed in order to decrease inflammation and provide a better clinical outcome to the patient.

DETAILED DESCRIPTION:
This study aims to compare effectiveness of the treatment with intra-articular administration of collagen-PVP versus hylan GF 20, using the International Knee Documentation Committee (IKDC) score, 6 months after treatment. Hypothesis to test is: If effectiveness of intra-articular collagen-PVP is not lower than hylan GF 20 treatment in knee osteoarthritis subjects, then, statistically significant difference would not exist in IKDC score mean increase among treatment groups, after six months.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 40 and 80 years old
* Osteoarthritis in the knee rated II or III (Kellgren-Lawrence Grading Scale).
* Pain intensity (MOS Pain Severity Scale) greater than 40.
* Subject able to understand, co-operative and reliable.
* Written informed consent.

Exclusion Criteria:

* Acute arthritis in the knee.
* Ongoing anticoagulant therapy.
* Skin infection at the injection site.
* Systemic or intraarticular (target knee) corticosteroids in the past 3 months.
* Viscosupplementation (target knee) in the past year
* Arthroscopy/osteotomy/surgery in the past 5 months (target knee).
* Any surgery scheduled in the next 6 months
* Concomitant rheumatic disease (rheumatoid arthritis, spondyloarthritis, systemic lupus erythematosus, fibromyalgia).
* Severe varus/valgus deformity (>15°).
* Frontal deformity greater than 20 degrees
* History of allergy or hypersensitivity to hyaluronic acid or avian proteins
* History/present evidence of: metabolic joint diseases; crystal arthropaties; ochronosis; acromegaly; haemochromatosis; Wilson's disease; primary osteochondromatosis; heritable disorders.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-08-01 (Estimated); Primary Completion 2021-02-28 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
International Knee Documentation Committee (IKDC). | Evaluation will be conducted at Baseline and 6 months after first infiltration
  Change from Baseline in International Knee Documentation Committee (IKDC) subjective score at 6 months. The IKDC subjetive form is a patient-reported outcome, which contains sections on knee symptoms (7 items), function (2 items), and sports activities (2 items).The IKDC is scored by summing the scores for the individual items and then transforming the score to a scale that ranges from 0 to 100 (add the score for each item and divide by the maximum possible). The transformed score is interpreted as a measure of function such that higher scores represent higher levels of function and lower levels of symptoms. A score of 100 is interpreted to mean no limitation with activities of daily living or sports activities and the absence of symptoms.

SECONDARY OUTCOMES:
Change in Pain Intensity | Evaluation will be conducted at Baseline, 2 months, 3 months and 6 months after first infiltration
  Change from Baseline in Pain Intensity score (MOS Pain severity scale) at 6 months. The Medical Outcomes Study (MOS) Pain Severity Scale is a 5-item scale to assess pain intensity (average and at the most), frequency, and duration over the last 7 days. Scores range from 0-100; higher score indicates more pain
Change in quality of life: EQS-5D | Evaluation will be conducted at Baseline, 2 months, 3 months and 6 months after first infiltration
  Change from Baseline in quality of life (EQS-5D) score at 6 months.
Changes in Urine Collagen Type II C-telopeptide Fragments | Evaluation will be conducted at Baseline, and 6 months after first infiltration
  Changes from baseline in Urine Collagen Type II C-telopeptide Fragments (uCTX-II) at 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Gabriel Horta Baas, Mérida, Yucatán, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Furuzawa-Carballeda J, Munoz-Chable OA, Barrios-Payan J, Hernandez-Pando R. Effect of polymerized-type I collagen in knee osteoarthritis. I. In vitro study. Eur J Clin Invest. 2009 Jul;39(7):591-7. doi: 10.1111/j.1365-2362.2009.02154.x. PMID 19453649
- [Background] Furuzawa-Carballeda J, Munoz-Chable OA, Macias-Hernandez SI, Agualimpia-Janning A. Effect of polymerized-type I collagen in knee osteoarthritis. II. In vivo study. Eur J Clin Invest. 2009 Jul;39(7):598-606. doi: 10.1111/j.1365-2362.2009.02144.x. Epub 2009 Apr 23. PMID 19397687
- [Background] Furuzawa-Carballeda J, Lima G, Llorente L, Nunez-Alvarez C, Ruiz-Ordaz BH, Echevarria-Zuno S, Hernandez-Cuevas V. Polymerized-type I collagen downregulates inflammation and improves clinical outcomes in patients with symptomatic knee osteoarthritis following arthroscopic lavage: a randomized, double-blind, and placebo-controlled clinical trial. ScientificWorldJournal. 2012;2012:342854. doi: 10.1100/2012/342854. Epub 2012 Apr 1. PMID 22545014